CLINICAL TRIAL: NCT02824575
Title: Phase Ib Study of Rebastinib Plus Antitubulin Therapy With Paclitaxel or Eribulin in Patients With Metastatic Breast Cancer
Brief Title: Rebastinib Plus Antitubulin Therapy With Paclitaxel or Eribulin in Metastatic Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Unfortunately, Deciphera management decided to not move forward with the rebastinib program and are terminating early.
Sponsor: Montefiore Medical Center (Other)
Collaborators: Deciphera Pharmaceuticals, LLC (Industry); Albert Einstein College of Medicine (Other)
Responsible Party: Principal Investigator, Jesus Anampa Mesias, Assistant Professor of Medicine, Montefiore Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016-6488
Record Dates: First submitted 2016-06-28; First posted 2016-07-06 (Estimated); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Breast Cancer; Breast Adenocarcinoma; Human Epidermal Growth Factor 2 Negative Carcinoma of Breast; Recurrent Breast Carcinoma; Stage IV Breast Cancer
Keywords: breast cancer; chemotherapy; metastasis; tumor micro-environment
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — rebastinib; DCC-2036; Paclitaxel; eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A1-2: Paclitaxel plus Rebastinib. (Experimental): * Arm A1 (Dose Escalation Cohort): Paclitaxel 80 mg/m2 weekly x 12 weeks plus Rebastinib (50 mg PO BID or 100 mg PO BID) beginning on cycle 1, day 1 and given continuously.
  * Arm A2 (Expansion Cohort): Paclitaxel 80 mg/m2 weekly x 12 weeks. Patients will be randomized to receive Rebastinib (at RP2D) beginning on cycle 1, day 1 OR cycle 2, day 1.
  Interventions: Drug: Rebastinib; Drug: Paclitaxel
- Arm B1-2: Eribulin plus Rebastinib. (Experimental): * Arm B1 (Dose Escalation Cohort): Eribulin Mesylate 1.4 mg/m2 day 1 & 8 q21 days plus Rebastinib (50 mg PO BID or 100 mg PO BID) beginning on cycle 1, day 1 and given continuously.
  * Arm B2 (Expansion Cohort): Eribulin Mesylate 1.4 mg/m2 day 1 & 8 q21 days. Patients will be randomized to receive Rebastinib (at RP2D) beginning on cycle 1, day 1 OR cycle 2, day 1.
  Interventions: Drug: Rebastinib; Drug: Eribulin Mesylate

INTERVENTIONS:
Drug: Rebastinib — 50 mg or 100 mg po BID continuously. Cycle duration: 21 days. Number of Cycles: 4 cycles or until progression or unacceptable toxicity develops.
  Other Names: DCC-2036
Drug: Paclitaxel — Paclitaxel 80 mg/m2 weekly. Cycle duration = 21 days. Number of Cycles: 4 cycles or until progression or unacceptable toxicity develops.
  Other Names: Taxol
  Arms: Arm A1-2: Paclitaxel plus Rebastinib.
Drug: Eribulin Mesylate — Eribulin 1.4 mg/m2 day 1 & 8. Cycle duration : 21 days. Number of Cycles: 4 cycles or until progression or unacceptable toxicity develops.
  Other Names: Halaven
  Arms: Arm B1-2: Eribulin plus Rebastinib.

SUMMARY:
The purpose of this study is to determine the safety and tolerability of rebastinib when combined with antitubulin therapy with paclitaxel or eribulin in patients with advanced breast cancer.

DETAILED DESCRIPTION:
Metastasis is the primary cause of death from breast cancer, invasive carcinoma cells in mouse and rat mammary tumors co-migrate accompanied by macrophages towards intravasation sites . The intravasation occurs at sites where a TIE2-expressing macrophage, a mena-expressing tumor cell, and an endothelial cell are in direct contact, forming a micro-anatomic structure called tumor micro-environment of metastasis (TMEM). Ablation of the presence or activity of the TMEM associated macrophages blocks intravasation at TMEM demonstrating an essential role of perivascular macrophages in TMEM function. Rebastinib, a TIE2 inhibitor , blocks TMEM assembly and function in-vivo and in-vitro assays. We hypothesize that rebastinib combined with antitubulin therapy (eribulin or paclitaxel) could improve clinical outcomes in breast cancer by preventing intravasation at TMEM sites and preventing further metastasis.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of the breast that is HER2 (human epidermal growth factor receptor 2) negative; based on ASCO(american society of clinical oncology)/ CAP (college of American Pathologists) guidelines as: (a) IHC (immuno-histochemistry) 1+ negative or IHC 0 negative; or (b) ISH (in situ hybridization ) negative using single probe ISH( average HER2 copy number < 4.0 signals/cell), or dual probe ISH ( HER2/CEP17 ratio <2.0, average HER2 copy number <4.0 signals/cell)
2. Metastatic breast cancer not amenable to potentially curative surgery. Patients must have disease that is measurable and/or non-measurable as defined by RECIST 1.1 criteria
3. Prior chemotherapy and/or endocrine therapy. Patients will be assigned to arm A or arm B depending on their prior exposure to paclitaxel and eribulin.

   * Arm A: Rebastinib plus paclitaxel: Up to two prior non-taxane chemotherapy regimens for metastatic or incurable locally advanced disease permitted (no prior paclitaxel, docetaxel, or eribulin for metastatic disease)..Prior therapy with paclitaxel or docetaxel in the neo/adjuvant setting is allowable if there is at least a 6 month interval between the last adjuvant/neoadjuvant paclitaxel or docetaxel dose and recurrence.
   * Arm B: Rebastinib plus Eribulin: Patients must have previously received at least two chemotherapeutic regimens for the treatment of metastatic disease (no prior eribulin, but prior paclitaxel, nab-paclitaxel, or docetaxel allowed). Prior therapy should have included a taxane in either the adjuvant or metastatic setting.
   * Arms A and B: Patients with hormone receptor positive disease must have had progressive disease and at least 2 lines of endocrine therapy, including one endocrine regimen used in combination with an approved CDK 4/6 (cyclin-dependent kinase ) inhibitor (eg, palbociclib). Relapse while receiving or within 6 months of completing adjuvant endocrine therapy may be considered failure of one prior endocrine regimen
4. Female and age >18 years. Because breast carcinoma is a disease of adults that rarely occurs in children, children are excluded from this study. In addition, the safety of rebastinib in pediatric patients has not been evaluated.
5. ECOG (Eastern Cooperative Oncology Group) performance status 0 or 1.
6. Normal organ and marrow function as defined below within 2 weeks of registration (except where specified otherwise):

   Leukocytes >3,000/µL ; Absolute neutrophil count >1,500/µL ; Platelets >100,000/ µL Hemoglobin > 9 g/dL ; Total bilirubin (within normal institutional limits) AST (aspartate aminotransferase)/ALT (alanine aminotransferase) <2.5 X institutional upper limit of normal ; Creatinine (within normal institutional limits) ; EKG QTc < 450 msec (females)

   Left ventricular ejection fraction at or above institutional lower limits of normal (by echocardiogram within 12 weeks of registration) ; Glucose (within normal limits) Serum calcium & phosphorus (within normal institutional limits); Negative urine or serum B-HCG(Beta-Human Chorionic Gonadotropin)
7. No significant ocular disease: No prior known history of retinal neovascularization, macular edema or macular degeneration. Patients without such a history are required to have a baseline ophthalmologic exam as part of screening, and must not have evidence of retinal neovascularization, macular edema or macular degeneration on the screening exam in order to be eligible.
8. No other active cancer: Patients must be disease-free of prior invasive malignancies for > 2 years with the exception of curatively-treated basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix. Patient with the following prior or concurrent diagnoses are eligible: lobular carcinoma in situ, contralateral ductal carcinoma in situ, or contralateral invasive ductal and/or lobular carcinoma.
9. Women of child-bearing potential must not be pregnant or breast feeding. They must also agree to use adequate contraception (hormonal or barrier method of birth control) and not be breast feeding prior to study entry, for the duration of study participation, and for up to 30 days after completion of all protocol therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study or up to 30 days after completion of protocol therapy, she should inform her treating physician immediately.
10. Ability to understand and the willingness to sign a written informed consent document.
11. At least 30 days from major surgery before study enrollment, with full recovery.
12. Concomitant therapy with bisphosphonates, RANKL inhibitors or growth-colony-stimulating factor (G-CSF) is allowed as per physician decision.
13. Expansion cohort: Patients for the expansion cohort must have a CTC (TelomeScan) drawn in the screening phase if other eligibility criteria are met, and must be CTC-positive in order to be eligible for enrollment in the expansion cohort.

Exclusion Criteria:

1. History of allergic reactions attributed to compounds of similar chemical or biologic composition to Rebastinib or other agents used in the study (e.g., Cremophor)
2. History of cardiac disease, including: (a) myocardial infarction within 6 months of the start of study, (b) history of QTc(corrected QT interval ) prolongation or QTc >/= 450 msec on screening EKG, history of additional risk factors for Torsade de pointes( e.g., heart failure, hyperkalemia, and family history of long QT syndrome. (c) Use of concomitant drugs that prolong QT/QTc interval.(see "Study reference manual" for further details) (d) New York Heart Association class III or IV heart disease, (e), active ischemia or any other uncontrolled cardiac condition such as angina pectoris, clinically significant cardiac arrhythmia requiring therapy.
3. bIntercurrent illness that would substantially increase the risk of treatment associated complications (e.g., active infection, uncontrolled diabetes mellitus or hypertension) and/or psychiatric illness/social situations that would interfere with the patient's ability to comply with the treatment regimen.
4. Patients with HIV infection are excluded from the study because of possible pharmacokinetic interactions with Rebastinib and antiretroviral therapy.
5. Patients with untreated brain metastasis are excluded. Patients with a prior history of brain metastasis are eligible if they have received prior brain radiation, have improved or stable intracranial disease for at least 3 months after completion of last course of radiation, and are not taking corticosteroids for treatment of brain metastasis. Patients with a prior history of brain metastases who meet other eligibility criteria
6. Treatment with other chemotherapy regimen within the past 2 weeks.
7. Treatment with trastuzumab, bevacizumab or other targeted therapies within the past 4 weeks.
8. Patients who have not recovered (i.e., CTCAE Grade ≤1 or baseline) from an adverse event due to a previously administered agent, excluding alopecia.
9. Patients with Grade >1 neuropathy
10. Patients with uncontrolled hypertension (defined as systolic blood pressure > 150 and/or diastolic blood pressure > 90 mm/mg).
11. Patients that have a malabsorption syndrome or other illness which could affect oral absorption

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-07; Primary Completion 2021-12-27 (Actual); Study Completion 2021-12-27 (Actual)

PRIMARY OUTCOMES:
Recommended Phase 2 dose(RP2D). | After 1 treatment cycle (3 weeks) during dose escalation cohort (N=24)
  Arm A: To determine the recommended phase II dose (Arm A1 - dose escalation cohort) and overall safety profile (Arm A2 - expansion cohort) of Rebastinib (50 mg PO BID or 100 mg PO BID) given concurrently with weekly paclitaxel (80 mg/m2 weekly x 12 ) over 3 consecutive weeks (1 cycle) in patients with metastatic breast cancer.
  Arm B: To determine the recommended phase II dose (Arm B1 - dose escalation cohort) and overall safety profile (Arm B2 - expansion cohort) of Rebastinib (50 mg PO BID or 100 mg PO BID) given concurrently with weekly eribulin (1.4 mg/m2 days 1 and 8 every 21 days) over 3 consecutive weeks (1 cycle) in patients with metastatic breast cancer.

SECONDARY OUTCOMES:
Median Progression Free Survival (PFS) | From treatment start until progression or death, whichever occurs first, assessed up to 36 months
  Arm A1-2 and Arm B1-2 (evaluate separately for each arm): To determine the progression-free survival of patients treated with Rebastinib plus paclitaxel, and Rebastinib plus eribulin (at all Rebastinib dose levels).
Median Overall Survival (OS). | From treatment start until death by any cause, assessed up to 36 months.
  Arm A1-2 and Arm B1-2 (evaluate separately for each arm): To determine overall survival of patients treated with Rebastinib plus paclitaxel, and Rebastinib plus eribulin (at all Rebastinib dose levels).
Clinical benefit rate | Proportion of patients who achieved complete response or partial response for at least 24 weeks after study start.
  Arm A1-2 and Arm B1-2 (evaluate separately for each arm): To determine clinical benefit rate of patients treated with Rebastinib plus paclitaxel, and Rebastinib plus eribulin (at all Rebastinib dose levels).
Change of ANG1 and ANG2 levels | Before and after cycle 1( week 3) for each patient.
  Arm A1-2 plus Arm B1-2 (evaluate combined dataset including both arms): To determine correlation between Rebastinib and angiopoietin (ANG1 and/or ANG2) levels (a surrogate marker for TIE2 inhibition)
Change in Circulating Tumor Cells (CTC) levels. | Before and after cycle 1( week 3) for each patient.
  Arm A2 plus Arm B2: To perform an exploratory analysis of the effects of Rebastinib plus antitubulin therapy on circulating tumor cell (CTCs) during cycle 1, by comparing CTCs during cycle 1 in patients randomized to receive or not rebastinib during cycle 1.
Change in TIE-2 expressing monocyte levels. | Before and after cycle 1( week 3) for each patient.
  Arm A2 plus Arm B2: To perform an exploratory analysis of the effects of Rebastinib plus antitubulin therapy on TIE-2 expressing monocytes (TEM) during cycle 1.
Change in TMEM score. | Before and after cycle 1( week 3) for each patient.
  Arm A2 or Arm B2: To perform an exploratory analysis of the effects of Rebastinib plus antitubulin therapy on TMEM score and TMEM function in a cohort of up to 6 patients with metastatic cancer who have their primary tumor in place and are agreeable to up to 2 research biopsies of the primary tumor before and during (i.e., after 3 weeks of) Rebastinib therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Jesus D Anampa Mesias, M.D, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No